CLINICAL TRIAL: NCT00940992
Title: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Dose-Range Study of DER 45 EV Gel, 1% and 5%, and Vehicle Gel in the Treatment of Rosacea
Brief Title: A Study of DER 45-EV Gel to Treat Rosacea
Acronym: SGTDER45EV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SGT DER 45 EV 09
Record Dates: First submitted 2009-07-14; First posted 2009-07-17 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2014-12

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DER 45 EV Gel, 1% (Experimental): DER 45 EV Gel, 1% topically applied once daily to face for 12 weeks
  Interventions: Drug: DER 45 EV
- Vehicle (Placebo Comparator): Placebo Gel applied topically once a day for 12 weeks
  Interventions: Drug: Vehicle
- DER 45 EV Gel, 5% (Experimental): DER 45 EV Gel, 5% applied topically once a day for 12 weeks
  Interventions: Drug: DER 45 EV

INTERVENTIONS:
Drug: DER 45 EV — Topical application to face for 12 weeks
  Arms: DER 45 EV Gel, 1%; DER 45 EV Gel, 5%
Drug: Vehicle — Topical application to face for 12 weeks
  Arms: Vehicle

SUMMARY:
To identify lowest efficacious dose of DER 45 EV Gel, 1% and 5% verses vehicle in patients with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age or older
* Facial rosacea, with 12 or more inflammatory lesions (with no more than 2 nodules)
* Mild, Moderate or Severe (2, 3 or 4) rating of rosacea on the IGA
* Females of child-bearing potential must have negative urine pregnancy test result at baseline and must be willing to use an effective form of contraception throughout the study

Exclusion Criteria:

* Subjects who are pregnant, breast feeding, or planning a pregnancy during the study
* Allergy or sensitivity to ingredients in test product
* Any dermatological conditions of the face that may interfere with study evaluations
* Subjects unable to avoid or minimize exposure to factors that may exacerbate or trigger rosacea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Levy-Hacham, PhD, Study Director — Sponsor GmbH
Locations (10):
- United States (10):
  - Baumann Cosmetic & Research Institute, Miami, Florida
  - FXM Research Corp, Miami, Florida
  - Augusta Centre for Dermatology and Skin, Augusta, Georgia
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Search of Rochester, Inc, Rochester, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc, Austin, Texas
  - J & S Studies, Inc, College Station, Texas
  - Premier Clinical Research, Spokane, Washington
  - Madison Skin and Research, Inc, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DER 45 EV Gel, 1% | Vehicle | DER 45 EV Gel, 5%
Started | 32 | 30 | 30
Completed | 28 | 28 | 28
Not Completed | 4 | 2 | 2
Not completed — Adverse Event | 2 | 0 | 1
Not completed — subject request | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DER 45 EV Gel, 1% | Vehicle | DER 45 EV Gel, 5% | Total
Number analyzed (Participants) | 32 | 30 | 30 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.50) | 50.5 (12.56) | 52.2 (12.66) | 51.2 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 23 | 67
  Male | 10 | 8 | 7 | 25
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 30 | 92
number of inflammatory lesions [Mean (Standard Deviation); unit: number of inflammatory lesion] — minimum of 12 inflammatory lesions
  number of inflammatory lesion | 28.6 (27.76) | 19.9 (8.64) | 22.9 (16.89) | 23.9 (19.76)

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (IGA) Improvement From Baseline
Description: The proportions of subjects with the primary measure of success at week 12 /end of study ,defined as a 2-grade improvement in the IGA (Investigator Global Assessment) relative to Baseline. The Investigator Global Assessment grades are: Grade 0 (Clear), Grade 1 (Almost Clear), Grade 2 (Mild), Grade 3 (Moderate) and Grade 4 (Severe).
Time Frame: Baseline to Week 12 / end of treatment
Measure: Number; unit: percentage of subjects
Arm/Group | DER 45 EV Gel, 1% | Vehicle | DER 45 EV Gel, 5%
Number analyzed (Participants) | 32 | 30 | 30
percentage of subjects | 37.5 | 20.0 | 53.3

2. Primary Outcome: Change in Inflammatory Lesion Counts From Baseline
Description: The LS mean changes from Baseline in inflammatory lesion count at Week 12.
Time Frame: Baseline to Week 12 / end of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: Inflammatory lesions
Arm/Group | DER 45 EV Gel, 1% | Vehicle | DER 45 EV Gel, 5%
Number analyzed (Participants) | 32 | 30 | 30
Inflammatory lesions | -21.5 [-27.5 to -15.4] | -8.8 [-15.1 to -2.5] | -14.7 [-21.0 to -8.4]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | DER 45 EV Gel, 1% | Vehicle | DER 45 EV Gel, 5%
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 7/32 | 11/30 | 7/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DER 45 EV Gel, 1% (N=32) | Vehicle (N=30) | DER 45 EV Gel, 5% (N=30)
Application site dermatitis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site reaction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Cyst (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other